CLINICAL TRIAL: NCT00741455
Title: Non-Myeloablative Chemotherapy Followed by HLA-Matched Related Allogeneic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Chemotherapy Followed by Allogeneic Stem Cell Transplantation for Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John M. Hill, Jr., MD, Director, Allogeneic Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0345
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Hematologic Malignancies
Keywords: Non-myeloablative transplant; Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Multiple Myeloma; Non-Hodgkin's Lymphoma; Myelodysplastic syndrome; Chronic Lymphocytic Leukemia; Hodgkin's Disease
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease | interventions — Stem Cell Transplantation; Granulocyte Colony-Stimulating Factor; fludarabine; Cyclophosphamide; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Treatment (Experimental): Chemotherapy, stem cell transplantation, HLA-Matched related allogeneic stem cell transplantation, leukapheresis, G-CSF, peripheral blood stem cell transplant, fludarabine, cyclophosphamide, donor lymphocyte infusion, cyclosporine, methotrexate
  Interventions: Procedure: Stem Cell Transplant; Drug: G-CSF; Drug: Fludarabine; Drug: cyclophosphamide; Drug: Cyclosporine; Drug: Methotrexate

INTERVENTIONS:
Procedure: Stem Cell Transplant — Donor: Prior to mobilization, leukapheresis to collect CD3+ cells. The donor will then receive G-CSF (10 mcg/kg/day) with leukapheresis collection of peripheral blood stem cells on days 5, 6 and 7 as needed. Goal of leukapheresis will be > 5 x 106 CD34+cells/kg of recipient.
  Patient: Peripheral Blood Stem Cell (PBSC) Transplant. Fludarabine 25mg/m2/d IV over 30 minutes on days -6 to -2, followed by cyclophosphamide 1g/m2/d IV on days -3 and -2. This will be followed by allogeneic stem cell infusion 48 hours later.
  Donor Lymphocyte Infusion (DLI) and Adjustment of Immunosuppression: Cyclosporine (CSA) and methotrexate (MTX) will be used for GvHD prophylaxis with target CSA levels of 200-400 ng/ml.
  Other Names: HLA-Matched Related Allogeneic Stem Cell Transplantation
Drug: G-CSF — 10 mcg/kg/day on days 5, 6, and 7
Drug: Fludarabine — 25 mg/m2/d IV over 30 minutes on days -6 to -2
Drug: cyclophosphamide — 1 g/m2/d IV on days -3 and -2
Drug: Cyclosporine — used for GvHD prophylaxis with target CSA levels of 200-400 ng/ml
Drug: Methotrexate — used for GvHD prophylaxis with target CSA levels of 200-400 ng/ml

SUMMARY:
The purpose of this study is to determine disease-free survival, overall survival, time to progression, regimen-related toxicity and/or treatment-related mortality in patients with hematologic malignancies treated with non-myeloablative chemotherapy followed by allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Allogeneic bone marrow transplantation (BMT) became feasible in the 1960s after elucidation of the Human Leukocyte Antigen (HLA) complex. Since then, the therapy has evolved into an effective treatment for many hematologic disorders. Otherwise incurable malignancies are frequently cured by this approach, with the likelihood of cure ranging from 10% to 85%, depending on the disease and the disease status. The treatment strategy incorporates very large doses of chemotherapy and often radiation to eliminate cancer cells and to immunosuppress the recipient to allow the engraftment of donor cells. Donor cells give rise to hematopoiesis within two to three weeks, rescuing the patient from the effects of high dose therapy. In the ideal situation, immune recovery and recipient-specific tolerance occurs over the following 6-18 months, and the patient is cured of their underlying malignancy, off immunosuppression, with a functionally intact donor-derived immune system. However, complications are common and include fatal organ damage from the effects of high dose chemotherapy, infection, hemorrhage, and, in particular, graft-versus-host disease (GvHD). A realistic estimate of transplant-related mortality in the standard HLA-matched sibling setting is approximately 25%. The risk of treatment-related mortality limits the success and certainly precludes its use in older patients. Thus, new strategies in transplantation are needed.

With the growing understanding that much of the curative potential of allogeneic bone marrow or stem cell transplant (SCT) is from an immune anti-tumor effect of donor cells, known as graft-versus-leukemia (GvL) or graft-versus-tumor (GvT), a new strategy is being employed that shifts the emphasis from high-dose chemo-radiotherapy to donor-derived, immune-mediated anti-tumor therapy. In this approach, patients receive preparative regimens that, while having some anti-tumor activity, are mainly designed to be immunosuppressive enough to allow engraftment of donor stem cells and lymphocytes. Engrafted lymphocytes then mediate a GvL effect; if the GvL effect of the initial transplant is not sufficient, then additional lymphocytes may be infused (achievement of engraftment allows additional lymphocytes to "take" in the recipient without requiring any additional conditioning of the recipient). The lower intensity of the preparative regimen lessens the overall toxicity by minimizing the doses of chemo-radiotherapy. In addition, less intensive preparative regimens may be associated with less GvHD, as much evidence suggests that high-dose therapy contributes to the syndrome of GvHD by causing tissue damage, leading to a cytokine milieu which enhances activation of graft-versus-host (GvH) effector cells. Thus, such an approach may allow the safer use of allogeneic transplants in standard populations and may allow extension of allogeneic transplantation to patients who could not receive standard (myeloablative) transplants because of age or co-morbidities. This protocol investigates a non-myeloablative transplant approach, using fludarabine and cyclophosphamide, to allow engraftment of allogeneic cells, which may then mediate anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Diseases

  1. Chronic myelogenous leukemia (CML)

     * First chronic phase or later
     * Accelerated phase
  2. Acute myelogenous or lymphoblastic leukemia (AML or ALL)

     * Second or subsequent remission
     * Patients who have failed an autologous PBSC transplant
     * First remission with poor risk features, including, but not limited to: For AML- complex chromosome karyotype, abnormalities of chromosome 5 or 7, 12p-, 13+, 8+, t(9;22), t(11;23) For ALL- t(9;22), t(4;11), t(1;19), myeloid antigen coexpression
  3. Myelodysplastic syndrome (MDS)
  4. Multiple myeloma - high risk myeloma (poor responders, relapse after autologous PBSCT, chromosome 13 abnormalities)
  5. Hodgkin's disease

     * Primary refractory disease
     * Relapsed disease (first relapse or later)
     * Patients who have failed an autologous PBSC transplant
  6. Non-Hodgkin's lymphoma Low grade (by Working Formulation)

     * Relapsed, progressive disease after initial chemotherapy
     * Primary refractory disease or failure to respond (>PR) to initial chemotherapy
     * Patients who have failed an autologous PBSC transplant Intermediate grade (by Working Formulation)
     * Relapsed disease
     * Primary refractory disease or failure to respond (>PR) to initial chemo
     * Mantle cell lymphoma
     * Patients who have failed an autologous PBSC transplant
  7. Chronic lymphocytic leukemia (CLL)

     * Patients newly diagnosed with poor prognostic factors, including CD38 expression, Chromosome 11 or 17 abn
     * T-CLL/PLL
     * Relapsed or progressive disease, or refractory after Fludarabine
     * Patients who have failed an autologous PBSC transplant
* Donor Availability: Six of six matched HLA A, B and DR identical sibling (or parent or child) or 5/6 related donor with single mismatch at Class I antigen (A or B)
* Karnofsky performance status of >70%
* Serum bilirubin <2x upper limit of normal; transaminases <3x normal (unless due to disease)
* 24 hr urine creatinine clearance of >40 ml/min.
* DLCO >50% predicted
* Left ventricular ejection fraction >35%
* No active infection
* Non-pregnant female
* Signed informed consent
* No major organ dysfunction or psychological problems that preclude compliance and completion of the clinical trial.

Exclusion Criteria

* Major organ dysfunction
* Pregnant or lactating female
* Active infection
* Psychological problems that preclude compliance and completion of the clinical trial
* Any other condition, that in the judgement of the investigator, affects participant safety or overall participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-06; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Hill, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Kenneth R Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: Chemo, stem cell transplantation, HLA-Matched related allogeneic stem cell transplantation, leukapheresis, G-CSF, peripheral blood stem cell transplant, fludarabine, cyclophosphamide, donor lymphocyte infusion, cyclosporine, methotrexate
  Stem Cell Transplant: Donor: Prior to mobilization, leukapheresis to collect CD3+ cells. The donor will then receive G-CSF (10 mcg/kg/day) with leukapheresis collection of peripheral blood stem cells on days 5, 6 and 7 as needed. Goal of leukapheresis will be > 5 x 106 CD34+cells/kg of recipient.
  Patient: Peripheral Blood Stem Cell (PBSC) Transplant. Fludarabine 25mg/m2/d IV over 30 minutes on days -6 to -2, followed by cyclophosphamide 1g/m2/d IV on days -3 and -2. This will be followed by allogeneic stem cell infusion 48 hours later.
  Donor Lymphocyte Infusion (DLI) and Adjustment of Immunosuppression: Cyclosporine (CSA) and methotrexate (MTX) will be used for GvHD prophylaxis with target CSA levels of 200-400 ng/ml.
  G-CSF: 10 mcg/k
Period: Overall Study
Arm/Group | Study Treatment
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Bone Marrow Engraftment
Description: Rates of successful engraftment.
Time Frame: Within 30 days of bone marrow transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 17
Participants
  Engrafted </= 15 Days | 1
  Engrafted 16-30 Days | 15
  Engrafted >30 Days | 1

2. Secondary Outcome: Number of Participants Who Achieve Complete Donor Chimerism
Description: Complete donor chimerism
Time Frame: Post-transplant days +30, +60, +100, +180 and +365
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 17
Participants
  Complete Chimerism 30 Days Post Transplant | 2
  Complete Chimerism 60 Days Post Transplant | 2
  Complete Chimerism 100 Days Post Transplant | 3
  Complete Chimerism 180 Days Post Transplant | 3
  Complete Chimerism 365 Days Post Transplant | 4
  Chimerism Unknown | 1
  Did not achieve complete donor chimerism | 2

3. Secondary Outcome: Number of Participants Who Experienced Graft-Versus-Host-Disease
Description: Collect the number of incidents of acute and chronic graft-versus-host disease
Time Frame: Post-transplant procedure through death
Population: Data was not collected for this outcome measure
Arm/Group | Study Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival Measured in Participants
Description: Mortality rates in subjects after successful completion of a bone marrow transplant
Time Frame: Up to 15 Years Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 17
Participants
  Survival < 1 year post-transplant | 2
  Survival 1 to < 5 years post-transplant | 8
  Survival 5 to < 10 years post-transplant | 0
  Survival 10+ years post-transplant | 7

5. Secondary Outcome: Collection of Adverse Events
Description: Determine the level of toxicity experienced by subjects who receive protocol treatment and bone marrow transplant
Time Frame: Until the 6th Bone Marrow Transplant performed in subjects on study
Population: Data was not collected for this outcome measure
Arm/Group | Study Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Assess Disease Response
Description: Review and assess the tumor response rate
Time Frame: Post-transplant procedure through death
Population: Data was not collected for this outcome measure
Arm/Group | Study Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed for up to 15 years post-transplant. Adverse event data was not collected.
Description: Serious Adverse Event data was not collected. Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Study Treatment
All-Cause Mortality (participants affected / at risk) | 10/17
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT00741455/Prot_SAP_000.pdf